CLINICAL TRIAL: NCT01052389
Title: GiSAS Trial: Aripiprazole, Olanzapine, and Haloperidol in the Long Term Treatment of Schizophrenia.
Brief Title: Pragmatic RCT Comparing Aripiprazole, Olanzapine and Haloperidol in the Treatment of Schizophrenia
Acronym: GiSAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GiSAS 001; 2007-000278-22 (EudraCT Number)
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Pragmatic RCT; Aripiprazole; Olanzapine; Haloperidol; Metabolic syndrome; Drug discontinuation
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome | interventions — Aripiprazole; Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aripiprazole (Experimental): Aripiprazole (N05AX12)
  Interventions: Drug: Aripiprazole
- Olanzapine (Experimental): Olanzapine (N05AH03)
  Interventions: Drug: Olanzapine
- Haloperidol (Experimental): Haloperidol (N05AD01)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Aripiprazole — Patients allocated to aripiprazole will be prescribed daily oral dose of drug, based on individual response and side-effects. Suggested starting dose will be 10 mg/day and dose range will be 10-30 mg/day.
  Other Names: ATC code: N05AX12
  Arms: Aripiprazole
Drug: Olanzapine — Patients allocated to olanzapine will be prescribed daily oral dose of drug, based on individual patients' response and side-effect burden. Suggested starting dose will be 5 mg/day and dose range will be 10-20 mg/day.
  Other Names: ATC code: N05AH03
  Arms: Olanzapine
Drug: Haloperidol — Patients allocated to haloperidol FGA arm will be prescribed daily oral dose of drug, based on individual patients' response and side-effect burden.
  Suggested starting dose will be 1-3 mg/day and dose range 3-10 mg/day (chlorpromazine equivalents: suggested starting dose 50-100 mg/day; dose range 150-300 mg/day).
  Other Names: ATC code: N05AD01
  Arms: Haloperidol

SUMMARY:
The GiSAS study is a multi-centre randomized clinical trial that will involve about 80 italian community psychiatric services in Italy and will recruit 800 patients affected by schizophrenia.

In a sample of schizophrenic outpatients, it is hypothesized that there are significant differences in the overall tolerability and effectiveness of aripiprazole, olanzapine and haloperidol at 12 months.

It is a pragmatic trial. Thus, participants are selected to represent a broad range of "real-world" patients, all treatment medications are non-blinded and after randomization, the assigned drugs will be prescribed according to usual care practice.

The measure for effectiveness is retention of patients on the assigned treatment. The measure for tolerability is the onset of metabolic syndrome.

DETAILED DESCRIPTION:
Specific aim.

The GiSAS study is a randomized controlled superiority trial that aims to evaluate the tolerability and effectiveness of aripiprazole, olanzapine and haloperidol in outpatients with schizophrenia over a 12-month period.

Inclusion criteria.

* Age≥18.
* Patients entering the study must have a condition appropriate for changing the antipsychotic treatment or starting a new one.

Exclusion criteria.

* Diagnosis of metabolic syndrome.
* Diagnosis of diabetes mellitus type II.
* The patient has never been exposed to antipsychotic drugs.
* One of the studied treatments is clearly contraindicated.

Recruitment.

The study will be conducted in a broad array of clinical settings in order to provide generalizable and practically relevant study findings. The recruitment period will last 12 months in each participating center.

Study design.

The GiSAS study is a multi-centre RCT that will involve about 80 italian psychiatric services and will recruit 800 patients affected by schizophrenia.

In a non-selected sample of schizophrenic patients, it is hypothesized that there are significant differences in the overall safety, tolerability and acceptability of aripiprazole, olanzapine and haloperidol and consequently in their effectiveness.

It is a pragmatic trial. Thus, participants are selected to represent a broad range of "real-world" patients, including those with comorbid conditions (i.e. substance use disorders, medical problems.

Patients will be assessed:

* at baseline (all subjects);
* when monotherapy treatment is stopped;
* at 12 months (all subjects).

Pharmacological treatments.

In this study, the following drugs will be tested: (a) aripiprazole, (b) olanzapine, (c) haloperidol. All treatment medications are non-blinded.

After randomization, the assigned drugs will be prescribed according to usual care practice. Patients will be prescribed daily oral dose of the assigned drug, based on individual response and side-effects. For patients already taking an antipsychotic medication prior to study entry, tapering the previous medication over a period of four weeks will be allowed.

All the drugs used in each arm of GiSAS trial are currently licensed and marketed in Italy for the treatment of schizophrenia. No other antipsychotic medication will be allowed.

Concomitant psychotropic medication (e.g. benzodiazepines, antidepressants) and the use of non-psychotropic drugs will be allowed and routinely recorded.

Primary outcomes.

The measure for effectiveness is retention of patients on the assigned treatment at 12 months. The measure for tolerability is the onset of metabolic syndrome at 12 months (primary endpoint). Switching to another antipsychotic, adding a second antipsychotic or stopping antipsychotic treatment will be considered as drug discontinuation. Reasons for discontinuation will be registered and will be taken into account when creating the secondary outcomes.

In order to capture whether, when and why participants stop the assigned treatment or add concomitant medication, the patients' ongoing treatments will be monitored at least once a month.

The primary endpoint (i.e. Metabolic Syndrome) is assessed centrally by blinded independent observers.

All statistical analyses will be blinded and will include all randomized subjects following the intent-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* men and women, 18 years of age and over, who meet DSM-IV criteria for schizophrenia, based upon the Mini International Neuropsychiatric Interview;
* patients entering the study must, according to their own judgment in consultation with their physician, have a condition appropriate for (a) starting treatment with an oral antipsychotic medication or (b) changing antipsychotic treatment.

Exclusion Criteria:

* diagnosis of metabolic syndrome, defined as the fulfilling of at least 3 of the diagnostic criteria for the metabolic syndrome derived from Adult Treatment Protocol III (ATP III);
* diagnosis of diabetes mellitus type II;
* presence of an organic condition clearly contraindicating treatment with one of the studied drugs, e.g., pregnancy or breast-feeding;
* one of the studied treatments is positively known to be ineffective or not tolerable and consequently contraindicated;
* the patient has never been exposed to antipsychotic drugs;
* according to clinician's opinion, it is unlikely that the patient can be followed for the whole duration of the study (1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-07; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The measure for tolerability is the onset of metabolic syndrome as defined by meeting at least 3 of the following criteria: (1) abdominal obesity, (2) high triglycerides, (3) high HDL, (4) high blood pressure and (5) hyperglycaemia. | 12 months

SECONDARY OUTCOMES:
The primary measure for effectiveness is retention of patients on the assigned treatment at 12 months. Switching to another antipsychotic, adding a second antipsychotic or stopping antipsychotic treatment will be considered as drug discontinuation. | 12 months
  The trial takes account of two main outcomes, one for tolerability and one for effectiveness. Together, in fact, they must provide the most clinically relevant and convincing evidence directly related to the primary objective of the trial. The proportion of subjects who developed MS at one year was compared between the study groups and was adopted as primary endpoint. However, as the study design and conduction were focused on the one-year retention of the allocated monotherapy, the study power was estimated for this secondary endpoint too
Global functioning and symptomatology (GAF) | 12 months.
Time to discontinuation due to efficacy | 12 months.
Time to discontinuation due to side effects | 12 months
Worsening of metabolic profile | 12 months
  Defined as the onset of at least one metabolic syndrome criterion; onset of serum lipids abnormalities (dyslipidemia)
Neuroleptic side effects' self-rating (LUNSERS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Barbato, M.D., Principal Investigator — 'Mario Negri' Institute for Pharmacological Research; Alberto Parabiaghi, M.D., Study Director — 'Mario Negri' Institute for Pharmacological Research; Barbara D'Avanzo, Phil.D., Study Chair — 'Mario Negri' Institute for Pharmacological Research; Mauro Tettamanti, Biol.D., Study Chair — 'Mario Negri' Institute for Pharmacological Research
Locations (1):
- Department of Mental Health, Genoa, Liguria, Italy

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149
- [Derived] Ghio L, Natta W, Barbato A, Marcenaro M, Gotelli S, Jones PB, Parabiaghi A. Schizophrenia trial participation: perceived inclusion barriers and beliefs about antipsychotics. Pharmacopsychiatry. 2011 Jun;44(4):123-8. doi: 10.1055/s-0031-1277147. Epub 2011 Jun 27. PMID 21710401
- [Derived] Parabiaghi A, D'Avanzo B, Tettamanti M, Barbato A; GiSAS Study Group. The GiSAS study: rationale and design of a pragmatic randomized controlled trial on aripiprazole, olanzapine and haloperidol in the long-term treatment of schizophrenia. Contemp Clin Trials. 2011 Sep;32(5):675-84. doi: 10.1016/j.cct.2011.04.008. Epub 2011 Apr 30. PMID 21554991
- See also: GiSAS Study — http://gisas.marionegri.it
- See also: UE Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=gisas